CLINICAL TRIAL: NCT06194045
Title: A Randomized, Double-blinded Nutritional Study to Determine the Effect of a Concentrated Cetoleic Acid Fish Oil on Atopic Dermatitis
Brief Title: Nutritional Study to Determine the Effect of Fish Oil on Atopic Dermatitis
Acronym: CetoSkin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Møreforsking AS (Other)
Collaborators: Helse Møre og Romsdal HF (Other Government); Epax Norway AS (Industry); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 589440
Record Dates: First submitted 2023-12-05; First posted 2024-01-08 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis
Keywords: Cetoleic acid; LC-MUFA; Ezcema; Nutritional study
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Interventions are given as 1g bovine capsules of equal size, weight and appearance, and provided in identical bottles with a coded label.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC-MUFA oil (Experimental): 2x1g capsules containing concentrated marine oil from north atlantic fish
  Interventions: Dietary Supplement: LC-MUFA oil
- Placebo (Placebo Comparator): 2x1g capsules containing corn oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LC-MUFA oil — 2 x 1 g capsules containing marine oil from North Atlantic fish
  Arms: LC-MUFA oil
Dietary Supplement: Placebo — 2 x 1 g capsules containing corn oil
  Arms: Placebo

SUMMARY:
Atopic Dermatitis is associated with pronounced changes in the lipid composition in the skin. The lipid changes are influenced by and contributing to both the inflammatory circuit and the impaired barrier as well as changes in the skin microbiome This nutritional study will investigate the effect of long-chain monounsaturated fatty acid Cetoleic acid on atoptic dermatitis. Earlier studies have shown a anti-inflammatory effect of celoteic acid.

DETAILED DESCRIPTION:
Women and men will be recruited to a placebo or a cetoleic-rich fish oil group and be examined for the effect on atopic dermatitis before, during and after the study period.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 18-80 years of age.
* Diagnosed with active mild to moderate atopic dermatitis with an EASI of 1.1- 21.0.
* Willing to refrain from oil supplements (omega-3, borage, evening primrose, etc.) for 1 month before study begin (washout) and during the study
* Willing to take the study supplement for 6 months

Exclusion Criteria:

* Known allergy to fish products
* Subjects known to be pregnant or breast feeding
* Subjects perceiving systemically administered medication for AD (other than topical)
* Subjects with auto-immune diseases (except asthma and seasonal/perennial rhinitis)
* Subjects with a diagnosis of other skin diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
EASI | 6 months
  Change in EASI (Eczema Area and Serverity Index) POEM).
DQLI | 6 months
  Change in DQLI
POEM | 6 months
  Change in POEM (Patient Oriented Eczema Measure)
Itch Numerical Rating Scale (NRS) | 6 months
  Change in experienced itch on average the last 24 hours, and how the worst itch in the past 24 hours was. Scale from 0 (no itch) to 10 (worst imaginable itch).

SECONDARY OUTCOMES:
Fatty acid composition in red blood cells | 6 months
  Determine the change in fatty acid composition in red blood cells
Lipid compositions in skin | 6 months
  The change of ceramide/lipid composition in skin
Inflammation in skin | 6 months
  The change in inflammatory signalling molecules in skin
Blood lipids | 6 months
  The change in cholesterol/blood lipid profile
TEWL | 6 months
  The change in trans-epidermal water loss (TEWL)
Hydroxylated omega-3 fatty acids in plasma | 6 months
  The change of hydroxylated omega-3 fatty acids in plasma
Omega-3 index with EASI parameters | 6 months
  The association of omega-3 index with EASI parameters
Cetoleic acid with EASI parameters | 6 months
  The association of cetoleic acid content in RBCs with EASI parameters

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne Lihaug Hoff, Principal Investigator — Helse Møre og Romsdal HF
Locations (1):
- Helse Møre og Romsdal HF, Ålesund, Møre og Romsdal, Norway

IPD SHARING:
Plan to Share IPD: No
Data will be presented as collective statistical data.